CLINICAL TRIAL: NCT03324386
Title: HYPERTENSIVE PATIENT ADHERENCE TO TREATMENT: THE USE OF THERAPEUTIC COMMUNICATION ASSOCIATED WITH TECHNOLOGY EDUCATIONAL IN HEALTH PROMOTION"
Brief Title: The Use of Educational Technology in Improving Adherence Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Luiz Aparecido Bortolotto (Unknown); Chao Lung Wen (Unknown); Margarida Vieira (Unknown); Miriam Harume Tsunemi (Unknown); Isabela Ribeiro Braga Fistarol (Unknown); Jefferson Carlos de Oliveira (Unknown); Dante Marcelo Artiga Giorgi (Unknown); Heno Ferreira Lopes (Unknown); Fernanda Marciano Consolim-Colombo (Unknown); Ivonete Sanches Giacometti Kowalski (Unknown)
Responsible Party: Principal Investigator, Grazia Maria Guerra, Principal Investigator, InCor Heart Institute
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 08625112.7.0000.0068; 2012-50559-1 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2017-06-05; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Medication Nonadherence; Hypertension, Resistant to Conventional Therapy
Keywords: Hypertension; Tecnology; Nursing; Education
MeSH Terms: conditions — Medication Adherence; Hypertension Resistant to Conventional Therapy; Hypertension

STUDY DESIGN:
Intervention Model Description: VLE Group use the technology in a virtual learning environment(VLE) for distance learning (DL), HYBRID Group use the educational technology in the E-blended mode leraning, A Group he use of embracement strategy (relational strategies).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Individual Orientation: receiving individual orientation required by an embracement strategy characterized by 7 nursing visits at 20-day intervals, for 4 months);
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Individual Orientation (Experimental): This was a prospective randomized clinical study conducted with the following 4 groups of hypertensive patients: Experimental: individual orientation: receiving individual orientation required by an embracement strategy characterized by 7 nursing visits at 20-day intervals, for 4 months);The ntervention is composed by relational strategies characterized by interpersonal relationships
  Interventions: Behavioral: Experimental: Individual Orientation; Behavioral: Experimental: VLE for Distance Learning
- VLE for Distance Learning (Experimental): This was a prospective randomized clinical study conducted with the following 4 groups of hypertensive patients:Experimental: a technological education strategy for distance learning (DL), using a technological education strategy (E-Care of Hypertension) for Distance Learning (DL) characterized by 7 nursing visits at 20-day intervals, for 4 months). The intervention is composed by the use of equipment-oriented techniques or audio-visual aids in educational environments remotely accessed for health education specifically for hypertensive patients
  Interventions: Behavioral: Experimental: Individual Orientation; Behavioral: Experimental: E-blended Lerarning
- E-blended Learning (Experimental): This was a prospective randomized clinical study with the patient received experimental intervention: a technological education strategy with E-blended Learning modality with E-Care of Hypertension, associated with face-to-face consultation with the health professional and making 7 nursing visits at 20-day intervals, for 4 months. The intervention is composed by the use of equipment-oriented techniques or audio-visual aids in presential educational environments intended for health education specifically for hypertensive patients
  Interventions: Behavioral: Experimental: Individual Orientation; Behavioral: Experimental: VLE for Distance Learning; Behavioral: Experimental: E-blended Lerarning; Other: Conventional Therapy - Control Group
- No intervention (No Intervention): No type of intervention was performed making 2 nursing visits at baseline and 1 after 120 days (No intervention)

INTERVENTIONS:
Behavioral: Experimental: Individual Orientation — This approach may be individual orientation with by an embracement strategy (relational strategies) may be making 7 nursing visits at 20-day intervals, for 4 month.
  Arms: E-blended Learning; Individual Orientation; VLE for Distance Learning
Behavioral: Experimental: VLE for Distance Learning — Experimental: This approach may be associated with the use of educational technology (E-Care of Hypertension) in a virtual learning environment(VLE) for distance learning (DL) consultation with the health professional and making 7 nursing visits at 20-day intervals, for 4 months
  Arms: E-blended Learning; Individual Orientation
Behavioral: Experimental: E-blended Lerarning — This approach may be associated with the use of educational technology (E-Care of Hypertension) in the blended e-learning mode associated with face-to-face with the health professional and making 7 nursing visits at 20-day intervals, for 4 months
  Arms: E-blended Learning; VLE for Distance Learning
Other: Conventional Therapy - Control Group — This approach may be individual orientation with conventional therapy may be making 2 nursing visits at baseline and 1 after 120 days,
  Arms: E-blended Learning

SUMMARY:
Few studies show the benefits of educational technologies a support for the control of chronic diseases. The approach known as 'embracement' adopts relational strategies or soft technologies which promote bonding and may impact therapy adherence and quality of life in hypertensive patients.Objectives:To assess the impact of the embracement approach on therapy adherence, quality of life, and the white coat effect in hypertensive outpatients followed in a specialized clinic. This approach may be associated or not with the use of educational technology in a virtual learning environment(VLE) for distance learning (DL) and with use the educational technology in Blended E-learning (E-BLENDED)

DETAILED DESCRIPTION:
Hypertension (HBP) is an important risk factor for cardiovascular disease and has become a common public health problem world wide due to increased longevity. The challenge for next decades is to improve the adherence of patients with chronic degenerative diseases. It is detected that hypertension has been considered a risk factor for determining the incidence of cardiovascular diseases, which directs it to the high cost of treatment in Brazilian public health, therefore the prevention of impairment to health is a priority. Many patients with hypertension do not make the required behavioral changes in your lifestyle, do not forget to take medications or taking medication to fulfil the effective control of the disease. The present study aims to assess the impact of a health promotion program using the Therapeutic Communication and Educational Technology associated of the telemedicine (E-Care of Hypertension) in the performance improvement of patient adherence to treatment. This study aims to evaluation the impact of health promotion program on therapeutic compliance in hypertensive patients, of difficult control of blood pressure levels, with individual guidance through nursing consultation every 20 days, using the approach of "Therapeutic Communication" associated "Educational Technology" for a period of 120 days. For this study will be conducted with 60 patients randomly divided into four groups, according to the care of new cases registered in Ambulatory Hypertension Unit of Heart Institute at Medical School of São Paulo University. The sample will be selected for convenience in accordance with the established day of the week depending on availability of researchers and patients' consent. This approach may be associated or not with the use of educational technology in a virtual learning environment (VLE) for distance learning (DL).This was a prospective randomized clinical study conducted with the following 4 groups of hypertensive patients: This was a prospective randomized clinical study conducted with the following 4 groups of hypertensive patients: Embracement: Group receiving individual orientation required by an embracement strategy characterized by 7 nursing visits at 20-day intervals, for 4 months; Group VLE using a technological education strategy (E-Care of Hypertension) for distance learning (DL) and making 7 nursing visits at 20-day intervals, for 4 months; Control Group that performed 1 nursing visit at baseline and 1 after 120 days.). Group E-blended learning using a technological education strategy (E-Care of Hypertension) which is evaluating the influence of the use of educational technology associated with face-to-face consultation with the health professional (Blended E-learning) and making 7 nursing visits at 20-day intervals, for 4 months. At baseline and after 120 days, the following tools were applied: The Spielberger State-Trait Anxiety Inventory (STAI), the Morisky test, WHOQOL, and ambulatory blood pressure monitoring (ABPM). The VLE group had remote access to the "E-Care of Hypertension" site (6 specific educational modules).The E-BLENDED Group had acess to "E-Care of Hypertension" site (6 specific educational modules) with the presence of the nurse.

ELIGIBILITY:
Inclusion Criteria:

1. Have the medical diagnosis of arterial hypertension,
2. Have blood pressure levels equal or above 140 mmHg for systolic blood pressure (SBP), and equal or above 90 mmHg for diastolic blood pressure (DBP),
3. Must be able to swallow tablets and under drug treatment with antihypertensives,
4. Have digital accessibility through smart phones, tablets or notebooks and PCs.

Exclusion Criteria:

1. Patients with important cognitive impairment will be considered excluded, that is, with poor understanding of simple questions,
2. Clinical diagnosis of Alzheimer's disease, or chorea diseases that lead to cognitive impairment such as senile dementia,
3. Diagnosis of insulin dependent diabetes. -

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2015-04-25 (Actual); Study Completion 2017-02-17 (Actual)

PRIMARY OUTCOMES:
measure blood arterial pressure | 4 months
  At the first nurse interview (day 0: randomization), a questionnaire was used to obtain information related to general data, habits, history of disease, other risk factors for cardiovascular disease, and prescribed medications. This questionnaire was used only to characterize the adherence behavior and the risk factors at the beginning the study, but was not used to evaluate modifications of behavior during the study. Body weight and height were measured. Three consecutive measurements of BP were taken after the patient had rested for 5 min in the supine position.
Ambulatory Blood Pressure monitoring | 4 months
  Ambulatory BP monitoring was recorded at day ) in randomization and 120 days of follow-up for 24 h with a noninvasive ABPM (Space Labs 90207 monitor; Space Labs, Redmond, WA) with an appropriate-sized cuff. The monitor was placed on the nondominant arm and was set to take BP readings every 10 min during the day and every 20 min at nigh
Pill count | up to 4 months
  count of the compliments dispensed by the pharmacy and count of the empty blisters delivered in the consultation

SECONDARY OUTCOMES:
The brief version of the World Health Organization quality of life (WHOQOL-BREF) | 4 months
  Questinaire
The Duke University Religion Index (DUREL) for a brief measure of religiosity that can be included between religion and health outcomes. | 4 months
  the isntrument

IPD SHARING:
Plan to Share IPD: No